CLINICAL TRIAL: NCT00508794
Title: Biobehavioral Effects of Yoga During Breast Cancer Treatment
Brief Title: Effects of Yoga in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2005-0522; CA102385 (Other Grant/Funding Number: NCI); NCI-2010-00743 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-07-27; First posted 2007-07-30 (Estimated); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Tibetan Yoga; Stretching Program; Yoga; Quality of Life; Questionnaire; Survey
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 Yoga Program (Experimental): 3 sessions of yoga each week for 6 weeks. Questionnaire evaluating treatment-related symptoms during the middle of radiotherapy.
  Interventions: Behavioral: Yoga Group; Other: Questionnaire
- Group 2 Stretching Program (Experimental): 3 sessions of stretching each week for 6 weeks. Questionnaire evaluating treatment-related symptoms during the middle of radiotherapy.
  Interventions: Behavioral: Stretching Control Group; Other: Questionnaire
- Group 3 Waitlist Control Group (Other): Option of participating in the yoga or stretching program after the study has ended. Questionnaire evaluating treatment-related symptoms during the middle of radiotherapy.
  Interventions: Behavioral: Waitlist Control Group; Other: Questionnaire

INTERVENTIONS:
Behavioral: Yoga Group — 3 sessions of yoga each week for 6 weeks.
  Arms: Group 1 Yoga Program
Behavioral: Stretching Control Group — 3 sessions of stretching each week for 6 weeks
  Arms: Group 2 Stretching Program
Behavioral: Waitlist Control Group — Option of participating in the yoga or stretching program after the study has ended.
  Arms: Group 3 Waitlist Control Group
Other: Questionnaire — Questionnaire evaluating treatment-related symptoms during the middle of radiotherapy.
  Other Names: Survey

SUMMARY:
In this study researchers will examine the initial efficacy of implementing a yoga program for patients with breast cancer as an adjuvant to their radiotherapy. Patients with breast cancer who are undergoing radiotherapy will be randomly assigned to either a yoga group (YG), or a stretching (ST) control group, or a waitlist control (WL) group. Participants in YG and ST groups will attend three sessions each week throughout their 6-week radiotherapy schedule. The sessions will be coordinated with the treatment schedule and conducted adjacent to the treatment facility. Measures will be obtained prior to randomization, a brief assessment during the middle of radiation therapy, during the last week of radiation therapy, and 1, 3 and 6 months after the last radiation session. With the inclusion of two control groups in this randomized trial researchers will attempt to validate the benefits of yoga as an adjuvant to radiotherapy in patients with breast cancer wherein researchers will control for specific components of the yoga program and also examine some of the mechanisms that are necessary for the program to be effective.

Our specific aims in the proposed study are to:

* Conduct an initial evaluation of whether participation in the yoga program improves patients' fatigue and sleep disturbances. Fatigue and sleep will be assessed with self-report measures and the use of actigraphy for a more objective measure of sleep quality.
* Secondary end points will include examining QOL, mental health and objective physiological outcomes (blood samples for immune measures, saliva samples for cortisol levels, and heart rate variability).
* Exploratory analyses will examine some plausible mediators of the yoga program including cognitive processing, spirituality, and finding meaning in the cancer experience.

DETAILED DESCRIPTION:
If you choose to take part in this study, you will come to M. D. Anderson for your first visit. If this is not convenient, a researcher can visit you at your home. At this time, you will be asked to complete several questionnaires. The questions will ask about your sleeping habits, how you have been feeling, and your general QOL. This will take about 45-60 minutes to complete. Researchers, will then ask you to complete a daily sleep diary for the next 7 days. During this time, you will be given an actigraph watch to wear that will collect data about your day-time activity and sleeping habits. The watch should be worn 24 hours a day for 7 days a week. You will have an electrocardiogram (ECG - a test to measure the electrical activity of your heart) and your breathing rate will be measured.

After your first visit to M. D. Anderson or after a researcher has visited you at home, you will be randomly assigned (as in the toss of a coin) to one of 3 groups.

Participants in the first group will take part in a yoga program. If you are assigned to the yoga group, you will take part in 3 sessions of yoga each week for 6 weeks. You may take part in the yoga sessions any 3 days of the week. Each yoga session will last around 60 minutes. During the yoga sessions, you will also be asked to do breathing exercises and to perform different movements and meditation. None of the movements are difficult. You will be able to follow this program at your own pace.

Participants in the second group will take part in a stretching program. If you are assigned to the stretching group, you will take part in 3 sessions of stretching each week for 6 weeks. You may take part in the stretching sessions any 3 days of the week. Each stretching session will last around 60 minutes. During these stretching sessions you will be asked to do simple stretching exercises. None of the movements are difficult. You will be able to follow this program at your own pace.

Beginning with the second week, participants in the first and second groups will be asked to complete a brief questionnaire, about the yoga or stretching program, before the first class each week. The questionnaire will take about 1 to 2 minutes to complete. You will also have an ECG and your breathing rate will be measured before and after one of the classes during the third or fourth week and again during the last week. Each stretching and yoga session will be audio and video taped for the purpose of quality control.

Participants in the third group will not take part in the yoga or stretching program during this study. However, if you are assigned to this group, you will be given the option of participating in the yoga or stretching program after the study has ended. This will be after you have finished your last assessment.

All participants will complete a brief questionnaire during the middle of radiotherapy. The questionnaire will evaluate your treatment-related symptoms and will take about 15 minutes to complete.

During the last week of radiotherapy, and at 1, 3, and 6 months after the end of radiation treatment, all participants will be asked to fill out a packet of questionnaires (similar to those taken at the first visit). It should take about 45 minutes to complete all of the questionnaires. If it is not convenient for you to come to M. D. Anderson, a researcher can visit you at home to help with the questionnaires. You will then be asked to complete another daily sleep diary for another 7 days. During this time, you will wear an actigraph watch 24 hours a day for 7 days a week to collect the same data as before. During this time, you will have an ECG and your breathing rate will be measured.

All participants will be asked to refrain from participating in any other yoga classes for the duration of the study.

Your participation in this study will be over after your 6-month assessment.

This is an investigational study. Up to 180 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Women with Stage 0 - III breast cancer, undergoing daily adjuvant radiation for 6 weeks in the Department of Radiation Oncology at the M. D. Anderson
2. The participants will need to be 18 years of age or older.
3. Patients should be able to read, write, and speak English or Spanish.

Exclusion Criteria:

1. Patients who have a documented diagnosis of a formal thought disorder (e.g., schizophrenia) will be excluded from the study.
2. Patients with metastatic disease of the bone will be excluded to avoid any bone fractures that may result from yoga movements.
3. Patients with active/non-canalized deep vein thrombosis will be excluded from the study.
4. Patients who have not undergone any surgical treatment for their cancer will be excluded to ensure a more homogeneous sample.
5. Patients with extreme mobility issues (e.g., unable to get in and out of a chair unassisted) will be excluded.
6. Patients who have practiced yoga or taken yoga classes in the year prior to diagnosis will be excluded.
7. Patients diagnosed with lymphedema at baseline will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2006-03-09 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Fatigue and sleep assessed with self-report measures and actigraphy. | Measures will be obtained prior to randomization, a brief assessment during the middle of radiation therapy, during the last week of radiation therapy, and 1, 3 and 6 months after the last radiation session.

SECONDARY OUTCOMES:
To see if yoga will help to improve patients' quality of life (QOL) during treatment for cancer and during recovery from the effects of cancer treatment. | 4 Years
To learn if a yoga program is effective in helping to decrease emotional distress and improve physiological functioning. | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Cohen, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org